CLINICAL TRIAL: NCT04708626
Title: Epidemiology of Autoimmune Encephalitides and Paraneoplastic Neurological Syndromes in Sweden
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: DNR2019-03068
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Autoimmune Encephalitis; Paraneoplastic Neurological Syndrome
Keywords: autoimmune encephalitis; paraneoplastic neurological syndrome; neuronal antibody; epidemiology; incidence rate
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extended Cohort: Patients tested for any neuronal antibody in the Swedish population: All patients tested for any neuronal antibody in serum or CSF between 2015 and 2019 in Sweden.
  Interventions: Other: Description and analysis
- Core Cohort: Patients with a positive neuronal antibody test belonging to the Uppsala-Örebro region: All patients belonging to the Uppsala-Örebro health care region (a region in the middle of Sweden with a population of approximately 2.1 million), that tested positive for any neuronal antibody in serum or cerebrospinal fluid between 2015-2019.
  Interventions: Other: Description and analysis

INTERVENTIONS:
Other: Description and analysis — Collection of clinical, laboratory and radiological data from medical records.
  Groups: Core Cohort: Patients with a positive neuronal antibody test belonging to the Uppsala-Örebro region
Other: Description and analysis — Collection of laboratory data.
  Groups: Extended Cohort: Patients tested for any neuronal antibody in the Swedish population

SUMMARY:
Autoimmune encephalitis and paraneoplastic neurological syndromes are rare diseases caused by an abnormal immune response toward the nervous system. This can lead to life-threatening symptoms, but is in many cases treatable if a swift and correct diagnosis is made. Antibodies targeting neuronal proteins (i.e. "neuronal antibodies") can be detected in serum or cerebrospinal fluid (CSF) in about half of the patients suffering from these conditions. Although an important part of the diagnostical process of these conditions, diagnosis cannot be made only based on a positive antibody test, but the clinical findings have to be compatible as well. As these conditions are so rare, clinicians might struggle to interpret antibody test results.

In this study the investigators aim to estimate the incidence rate of autoimmune encephalitides and paraneoplastic neurological syndromes in the Uppsala-Örebro health care region in Sweden between the years 2015 and 2019. Medical records from patients belonging to the Uppsala-Örebro health care region (a region in the middle of Sweden with a population of approximately 2.1 million), that tested positive for any neuronal antibody in serum or CSF will be studied to obtain clinical, laboratory and radiological data. This data will be used to ascertain if diagnostic criteria are fulfilled as well as to describe clinical characteristics and identifying possible comorbidities.

DETAILED DESCRIPTION:
Methods:

1. Identification of extended cohort:

   The extended cohort consists of all patients in Sweden tested for any neuronal antibody in serum or CSF between 2015 and 2019. Patients will be identified by the only five laboratories that perform tests for neuronal antibodies in Sweden. The following neuronal antibodies will be included: AMPA 1 (Anti-Glutamate Receptor 1), AMPA 2 (Anti-Glutamate Receptor 2), Amphiphysin, CARP VIII (Carbonic Anhydrase-Related Protein VIII), CASPR2 (Contactin-associated protein-like 2), CV2/CRMP5 (collapsin response mediator protein 5), DPPX (dipeptidyl-peptidase-like protein 6), GABA B (γ-Aminobutyric acid-B receptor), GAD65 (glutamic acid decarboxylase) (>2000 IU/ml by ELISA in serum, or detected in CSF), glycine receptor, Homer 3, Hu (antineuronal nuclear antibody-type 1, ANNA-1), IgLON5 (immunoglobulin-like cell adhesion molecule 5 ), ITPR1 (inositol 1,4,5-trisphophate receptor type 1), LGI-1 (Leucine-rich glioma-inactivated 1), Ma2/Ta, NMDAR (anti-N-methyl-D-aspartate receptor), PCA-2 (Purkinje cell cytoplasmic antibody type 2), Tr (Trotter), Ri, SOX1(SRY-Box Transcription Factor 1), VGCC (Voltage-gated calcium channels), Yo, Zic4 (Zinc finger protein).
2. Identification of geographical region:

   Patients testing positive for any neuronal antibody in serum or CSF will be stratified according to which Swedish health care region that requested the test. Patients whose tests where requested by health care providers in the Uppsala-Örebro health care region (consisting of 7 smaller health care regions with a total population of approximately 2.1 million) will be selected.
3. Core cohort:

   Patients with a positive test result that belong to the Uppsala-Örebro health care region will be contacted and asked to participate in the study. Written informed consent must be signed to be included in the core cohort. If the patient is deceased, consent will be presumed.
4. Case ascertainment:

Medical records from patients included in the core cohort will be reviewed to obtain clinical, laboratory and radiological data. Ascertainment of a case is defined as the patient either fulfilling criteria of: 1) "definite PNS" according to Graus et. al 2021 or 2) "definite autoimmune limbic encephalitis" according to Graus et al. 2016 or 3) "definite anti-NMDA receptor encephalitis" according to Graus et al. 2016.

ELIGIBILITY:
Applicable only on Core Cohort:

Inclusion Criteria:

* All ages, both sexes.
* Neuronal antibody (AMPA 1, AMPA 2, Amphiphysin, CARP VIII, CASPR2, CV2/CRMP5, DPPX, GABA B, GAD65(>2000 IU/ml by ELISA in serum, or detected in CSF), glycine receptor, Homer 3, Hu, IgLON5, ITPR1, LGI-1, Ma2/Ta, NMDAR, PCA-2, Tr, Ri, SOX1, VGCC, Yo, Zic4), detected in serum or cerebrospinal fluid between 2015-2019
* Antibody test was requested by a health care facility in the Uppsala-Örebro health care region
* Signed informed consent. If the participant is deceased consent will be presumed

Exclusion Criteria:

* Incomplete personal data or social security number making it impossible to identify and/or contact the patient to get written consent
* Informed consent not signed. If the participant is deceased consent will be presumed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extended cohort: All patients in Sweden tested for any neuronal antibody (AMPA 1, AMPA 2, Amphiphysin, CARP VIII, CASPR2, CV2/CRMP5, DPPX, GABA B, GAD65 (>2000 IU/ml by ELISA in serum, or detected in CSF), glycine receptor, Homer 3, Hu, IgLON5, ITPR1, LGI-1, Ma2/Ta, NMDAR, PCA-2, Tr, Ri, SOX1, VGCC, Yo, Zic4), in serum or CSF between 2015 and 2019.
  Core cohort: All patients belonging to the Uppsala-Örebro health care region (a region in the middle of Sweden with a population of approximately 2.1 million), that tested positive for any neuronal antibody in serum or cerebrospinal fluid between 2015 and 2019. Patients will be identified by the only five laboratories that perform tests for neuronal antibodies in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of autoimmune encephalitides and paraneoplastic neurological syndromes in the Uppsala-Örebro health care region between 2015-2019 | 5 years
  Incidence rate of autoimmune encephalitides and paraneoplastic neurological syndromes in the Uppsala-Örebro health care region based on detection of neuronal antibodies in serum or CSF, with case ascertainment based on review of medical records and application of diagnostic criteria (Graus et al. 2016 and 2021).

SECONDARY OUTCOMES:
Positivity rate | 5 years
  Positivity rate - the number of positive tests divided by the number of total tests in the Swedish population for each year and for serum and CSF respectively.
False positivity rate | 5 years
  False positivity rate - the number of positive tests where case ascertainment fails divided by the total number of positive tests.
Estimated incidence rate of autoimmune encephalitides and paraneoplastic neurological syndromes in the Swedish population | 5 years
  Incidence rate of autoimmune encephalitides and paraneoplastic neurological syndromes in the Swedish population between 2015-2019 estimated from the incidence rates in the Uppsala-Örebro health care region as well as detection of neuronal antibodies in the entire Swedish population
Incidence rates of autoimmune encephalitides and paraneoplastic neurological syndromes | 5 years
  Yearly age-adjusted incidence rates for autoimmune encephalitides in the Uppsala-Örebro health care region between 2015-2019

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Burman, Assoc prof, Study Director — Uppsala University; Anna Rostedt Punga, Professor, Study Director — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided